CLINICAL TRIAL: NCT06193395
Title: Translation and Validation of the ICIQ-B in Danish Men and Women With Pelvic Floor Disorders
Brief Title: Translation and Validation of the ICIQ-B in Danish
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hanna Jangö (Other)
Responsible Party: Sponsor-Investigator, Hanna Jangö, MD, PhD, Associate Professor, Herlev Hospital
Organization: Herlev Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: VD-2020-04
Record Dates: First submitted 2023-12-06; First posted 2024-01-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2023-12

CONDITIONS: Anal Incontinence; Pelvic Floor Disorders; Quality of Life; Anal Sphincter Tear
MeSH Terms: conditions — Encopresis; Pelvic Floor Disorders | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients referred due to Pelvic Floor Disorders including anal incontinence (Experimental): all patients with PFDs are eligible
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — No intervention, only clinical testing of questionnaire

SUMMARY:
There are no validated scores in Danish revealing symptoms related to anal incontinence (AI). The International Consultation on Incontinence Questionnaire-Bowel (ICIQ-B) is an internationally recommended questionnaire that contains 21 items of which 17 are scored in three subscales: Bowel pattern; Bowel control and Quality of life. The aim was to translate and validate the ICIQ-B into Danish. The translation will be performed by a multidisciplinary team and the investigators will perform cognitive interviews and online testing of the questionnaire. The study only involves testing of a questionnaire and will not interfere with patient treatment.

DETAILED DESCRIPTION:
Background Anal incontinence (AI) is defined as the "complaint of involuntary loss of feces or flatus" and can significantly impact quality of life. Population studies have shown that 8-9% of adults suffer from AI with an equal distribution among men and women. There are different Patient Reported Outcome Measures (PROMs) regarding AI, but "the International Consultation on Incontinence Questionnaire Anal Incontinence Symptoms and Quality of Life Module" (ICIQ-B), first published in 2011, involved patients in the development of the questionnaire. The ICIQ-B is recommended by the International Consultation of Incontinence for both research and clinical use. There are no validated PROMs regarding AI in Danish, and therefore, the aim of this study was to translate and validate the ICIQ-B in Danish patients with pelvic floor disorders (PFD) with and without known AI.

Material and methods The ICIQ-B score contains 21 items and 17 of the 21 items are scored items. Each item is scored in an ordinal scale and each item contains a bother score rated on a numeric rank scale (NRS). The scored items are divided into three subscales covering: Bowel pattern (0-21), bowel control (0-28) and Quality of life (0-26) with a higher score indicating more symptoms.

We will recruit respondents from outpatient clinics in three hospitals in Denmark.

Inclusion criteria

* ≥ 18 years of age
* Fluency in Danish
* Referred to a pelvic floor clinic or to an outpatient clinic for a PFD or a routine follow-up

Exclusion criteria

• Cognitive disabilities that cause inability to complete a questionnaire

After translation of the questionnaire by an expert panel, the investigators will perform interviews, pretesting and test-retest. Healthcare professionals will inform patients about the study and hand out written patient information containing a QR-code and a weblink to access the questionnaire in REDCap (Research Electronic Data Capture). Informed consent will be given electronically. No physical examination will be performed as part of this study.

The hypotheses are that the ICIQ-B can discriminate between patients suffering from AI from patients without AI and that it will correlate moderately with a widely used AI score (St Marks score).

The investigators will evaluate content validity with floor and ceiling effect, structural validity of the three subscales, convergent validity (by correlating the ICIQ-B scores with the St. Marks score) and discriminant validity by comparing subscale scores between patients with and without known AI. The study will also evaluate reliability by evaluating internal consistency of the ICIQ-B subscales

Statistics Descriptive statistics will be used to show distribution of data about gender, age, and diagnoses. Analyses to compare groups will be performed using non-parametric statistical analyses. A level of significance with a p-value of ≤0.05 will be used. The analyses will be performed in SPSS.

Ethical considerations All participants will receive oral and written information about the study and sign an informed consent. Permission to perform the study is given from the Danish Data Protection Agency (VD-2020-04). The Regional Ethics committee confirmed that no permission from the committee was needed, since the study does not involve treatment of patients.

ELIGIBILITY:
Inclusion criteria

* ≥ 18 years of age
* Fluency in Danish
* Referred to a pelvic floor clinic or to an outpatient clinic for a pelvic floor disorder or a routine follow-up Exclusion criteria
* Cognitive disabilities that cause inability to complete a questionnaire

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 238 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Meaningful answers to single items and scores (ICIQ-B) in patients with and without anal incontinence and ability to discrimiante between groups of patients with and without anal incontinence | 15-30 minutes to complete the questionnaire (with or without interview-time included)
  translation into Danish

CONTACTS AND LOCATIONS:
Locations (1):
- Hanna Jangö, Herlev, Denmark

IPD SHARING:
Plan to Share IPD: No